CLINICAL TRIAL: NCT06091813
Title: Ambrosia: Evaluating the Effects of a Food-As-Medicine Platform on Gut Microbiome Composition and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Persephone Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PB-2023-01
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Impact of Dietary Chages Directed by Medical Nutrition Therapy on Gut Microbiome Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Directed Dietary Intervention (No Intervention): Control group without any directed dietary modifications
- Medical Nutrition Therapy (Experimental)
  Interventions: Behavioral: Nutrition Counseling

INTERVENTIONS:
Behavioral: Nutrition Counseling — Dietitian-led nutrition coaching via 5 Telenutrition visits, utilizing the Academy of Nutrition and Dietetics' Nutrition Care Process.
  Arms: Medical Nutrition Therapy

SUMMARY:
The objective of this study is to test whether dietary behavior modification impacts diet quality and stool microbiome composition and metabolism using microbial whole genome sequencing, targeted metabolomics, and immune profiling.

400 adults 18-64 years old at high risk for CRC (based on past colonoscopy findings or lifestyle risk factors) will be assigned to one of two cohorts, with approximately 200 participants in each.

* Cohort 1 will serve as the control group without any directed dietary modifications.
* Cohort 2 participants will receive medical nutrition therapy (MNT) via 5 Telenutrition (TN) visits with a registered dietitian (RD), utilizing the Academy of Nutrition and Dietetics' Nutrition Care Process.

Stool samples will be obtained for each subject at baseline and end of study. Whole genome sequencing, metabolite analysis, and immune profiling will be performed on the samples. Demographic data, general health information, diet and lifestyle information will be collected from the subjects (all self-reported). When applicable, notes from telenutrition appointments will also be collected. Diet information will be collected using the Picture Your Plate(TM) validated food questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 64 years old at the time of enrollment at high risk for colorectal cancer, defined as follows:

   1. EITHER a personal history of colorectal cancer, advanced adenoma, or 3 or more non-advanced adenomas in a single screening
   2. OR TWO of the following criteria:

      * One or more first-degree relatives with a history of colorectal cancer
      * Body mass index above 30 (Persephone will calculate given height and weight
      * Have smoked an average of 5 or more cigarettes (1/4 pack) per day for a continuous period of 10 years or more.
2. Able to provide stool samples at study start and after approximately 5 months
3. Willing and able to undergo virtual Medical Nutrition Therapy based on cohort assignment
4. Willing to complete online questionnaires concerning diet and lifestyle, in English
5. Competency in spoken and written English
6. Can provide written informed consent

Exclusion Criteria:

1. Subjects with known HIV, Hepatitis A, Hepatitis B, Hepatitis C
2. Known Familial Adenomatous Polyposis or Lynch Syndrome (aka Hereditary Non-Polyposis Colorectal Cancer or HNPCC) diagnosis
3. A history of Crohn's Disease, Inflammatory Bowel Disease, or chronic colitis.
4. Active cancer in the past 2 years, or currently undergoing any form of cancer therapy.
5. Confirmed case of COVID-19 or influenza within one month prior to enrollment
6. Oral or systemic antibiotic or probiotic use, or a known GI infection, within 3 months prior to enrollment
7. Engaged in a nutritional or dietary intervention in the past 3 months.
8. Women who are pregnant or plan to become pregnant in the next 6 months, or currently nursing.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 546 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Nutrition Counseling Microbiome Impact | 4 months
  Measure microbiome composition before and after 5 telenutrition visits by whole genome sequencing, and determine change in microbial composition as indicated by gUnifrac distance between the two datapoints.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Baum, MD, Principal Investigator — Independent
Locations (1):
- Persephone Biosciences, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to sign up for study — https://www.persephonebiosciences.com/ambrosia/